CLINICAL TRIAL: NCT01314144
Title: Does Continuous Wound Infusion of 0.2% Bupivacaine Provide Superior Analgesia Compared to Standard Opioid-based Therapy in Patients Following Axillary Clearance Surgery?
Brief Title: Use of Continuous Wound Infusion of Bupivacaine for Analgesia Following Axillary Clearance Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cork University Hospital (Other)
Responsible Party: Denise McCarthy, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-CUH
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: axillary clearance; wound infiltration; wound infusion; local anaesthetic wound infusion
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Experimental): Patients will receive intraoperative wound soakage with 20ml of 0.5% bupivacaine with adrenaline by the surgeon before closure and receive a continuous infusion of 4ml/hr of 0.2% bupivacaine delivered by an elastomeric pump the catheter of which will be placed by the surgeon in the wound before closure. Postoperative anlagesia will be provided with oxycodone, paracetamol and diclofenac.
  Interventions: Drug: Bupivacaine
- Control (No Intervention): Patients will receive morphine up to 0.1mg/kg intraoperatively. Postoperative analgesia will be provided with oxycodone, paracetamol and diclofenac.

INTERVENTIONS:
Drug: Bupivacaine — intraoperative wound soakage with 20ml of 0.5% bupivacaine with epinephrine and continuous infusion of 4ml/hr of 0.2% bupivacaine for 48 hours postoperatively
  Arms: Bupivacaine

SUMMARY:
Axillary clearance forms part of the surgical armamentarium for the treatment of breast cancer. Although the introduction of sentinel lymph node mapping and dissection has allowed for the decreased use of axillary clearance, it remains a frequently performed operation. Axillary clearance is associated with moderate postoperative pain.

We hypothesize that a continuous wound infusion of 0.2% Bupivacaine at 4ml/hr would provide superior analgesia, when compared to standard opioid-based analgesia, in patients undergoing axillary lymph node clearance surgery.

DETAILED DESCRIPTION:
The study will take the form of a prospective randomised clinical trial. The following assessment tools will be used

* The visual analogue scale (VAS) consists of a 100 mm horizontal line with the two end points labelled "no pain" and "worst pain ever". Patients are asked to mark on the line a point that corresponds to the level of pain intensity they feel. The score is obtained by measuring the distance (mm) from the left end of the line.
* The short-form McGill Pain Questionnaire (SF-MPQ) consists of 15 representative words from the sensory and affective categories of the standard McGill Pain Questionnaire. It also includes the present pain intensity and a VAS to provide overall indices of pain intensity. It has been shown to be sensitive to clinical changes brought about by various interventions, postoperative analgesic drugs (6).
* The Pain Catastrophising Score (PCS) is a 13 item instrument which asks patient to reflect on past painful experiences, and to indicate the degree to which they experienced each of these 13 thoughts or feelings, on 5-point scales with the end points; 0 = not at all, 4 = all the time. The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness (7).
* The Hospital Anxiety and Depression Score (HADS) is a 14-item scale, which screens for these, the two most common disturbances encountered in a medical setting (8).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing axillary clearance surgery
* ASA physical status I - III

Exclusion Criteria:

* Patient refusal
* Pre-existing pain conditions
* Regular use of opioid analgesia
* Pregnancy
* Severe cardiac, renal or hepatic disease
* Psychiatric illness precluding ability to give informed consent
* Intercurrent neurological disease
* Contraindications to bupivacaine or morphine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Pain on abducting the arm on the operative side to 90 degrees as measured using a 100mm visual analogue scale at 6 hours following surgery. | 6 hours postoperatively

SECONDARY OUTCOMES:
Pain (at rest and on movement) in the recovery room and at 6, 24 and 48 hours after surgery. | 48 hours postoperatively
Cumulative Oxycodone consumption at 6, 24 and 48 hours after surgery | 48 hours postoperatively
incidence of nausea and vomiting | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Denise M McCarthy, MB FCARCSI, Principal Investigator — Cork Universtiy Hospital
Locations (1):
- Cork Universtiy Hospital, Cork, Ireland